CLINICAL TRIAL: NCT05446389
Title: The Use of the Pacifier Activated Lullaby to Improve the Transition to Oral Feeding for Premature Infants With Chronic Lung Disease or Respiratory Distress Syndrome
Brief Title: PAL to Improve Oral Feeding for Infants With Chronic Lung Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution & the study was closed.
Sponsor: University of Missouri-Columbia (Other)
Collaborators: University of Georgia (Other)
Responsible Party: Principal Investigator, Emily Pivovarnik, Principal Investigator, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2091032
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lung Disease of Prematurity; Respiratory Distress Syndrome in Premature Infant; Bronchopulmonary Dysplasia; Preterm Birth
Keywords: Music Therapy; NICU; Pacifier Activated Lullaby; Premature Infant; Chronic Lung Disease; Oral Feeding
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Intervention Model Description: This study will utilize a clinical trial design. Participants will be randomized into two groups. One group will receive the PAL intervention, the other group serving as a no contact control. Participants will be matched based on sex, gestational age at birth, and neurologic injury. Infants in the intervention group will receive two PAL sessions a week until successfully transitioned to <2L of respiratory support and then receive one PAL session within 24 hours of their first oral feeding attempt.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Only one person (the primary investigator, who will be implementing the intervention) will be unmasked for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group (Experimental): Infants randomized in to the experimental group will receive the PAL intervention 2 times a week until the infant transitions to room air or < 2L high flow nasal cannula and is able to begin attempting feeds by mouth. The PAL is an FDA cleared medical device that has a sensor that will connect to the infant's pacifier and can read the infant's suck. Then, the device plays music as positive reinforcement to help improve sucking skills. This intervention typically lasts about 15 minutes and is implemented while the infant is receiving gavage feeds.
  Interventions: Device: Pacifier Activated Lullaby ®
- Control Group (No Intervention): Infants randomized in to the control group will not receive music therapy intervention throughout NICU admission.

INTERVENTIONS:
Device: Pacifier Activated Lullaby ® — Pacifier Activated Lullaby (PAL®) is a medical device that encourages and reinforces the development of non-nutritive sucking (NNS) of premature infants. This is accomplished by giving positive feedback in the form of music/mother's voice as an auditory input in direct response to effective sucking.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to investigate the effects of the Pacifier Activated Lullaby (PAL) intervention on the transition to oral feeding for preterm infants with chronic lung disease and respiratory distress syndrome that require non-invasive respiratory support at 34 weeks PMA. This study will utilize a clinical trial design. Participants will be randomized into two groups. One group will receive the PAL intervention, the other group serving as a no contact control. Participants will be matched based on sex, gestational age at birth, and neurologic injury. Infants in the intervention group will receive two PAL sessions a week until successfully transitioned to <2L of respiratory support and then receive one PAL session within 24 hours of their first oral feeding attempt.

DETAILED DESCRIPTION:
Infants in the Neonatal Intensive Care Unit at MU Healthcare receive consultations for music therapy services upon admission. The PAL intervention used in this study is a part of routine care that would happen regardless of participation in this study. The Music Therapist will discuss study with the parents of infants who meet inclusion criteria between 32 to 34 weeks PMA.

Clinical all infants on non-invasive respiratory support have a room air trial at 34 weeks PMA. Infants who fail their room air trail and are still on non-invasive respiratory support that is >2L will be randomized to either the control or intervention group. The control group will receive no additional intervention.

The experimental group will begin 2 PAL sessions per gestation week of age such that infants receive two sessions between 34 0/7 and 34 6/7, two sessions between 35 0/7 and 35 6/7, etc. When the infant is on <2L of respiratory support they will receive one more PAL session within 24 hours prior to their first oral feeding attempt.Infants in the experimental group will receive no additional PAL sessions after they begin oral feeding trials. PAL sessions will utilize the Pacifier Activated Lullaby device (PAL®) that is an FDA cleared medical device for use with preterm infants in the NICU. Sessions will be 15 minutes in length and be during the infant's gavage feed.The music therapist will get approval from the bedside RN prior to beginning any PAL sessions.The infant will be prompted with the pacifier by touching the pacifier to the infant's lips. If the infant doesn't accept pacifier in mouth after 3 attempts the music therapy will gently stroke the infant's cheeks to prompt the rooting reflex and then prompt with the pacifier. If the infant doesn't accept the pacifier in their mouth, then the music therapist will stop the session attempt and it will not count as a PAL session. If the infant pauses in non-nutritive sucking (NNS) for more than 30 seconds with music therapist will prompt the infant by moving pacifier in infant's mouth. This will be attempted 3 times if needed. If the infant still doesn't engage in NNS then the music therapy will stroke the infant's cheek and then move pacifier in mouth. This will be done twice. If the infant still does not engage in NNS then the session will be ended. The session will count if it lasted 8 minutes in length prior to the music therapist beginning prompting. If it was less than 8 minutes then it will not count towards a completed PAL session.

ELIGIBILITY:
Inclusion Criteria:

* All infants born less than 33 weeks PMA
* Infants enrolled prior to 35 weeks PMA
* Medically stable to tolerate minimal levels of auditory stimulation
* Approval from medical staff to begin intervention
* Requiring non-invasive respiratory support that inhibits the start of oral feeding, including: Continuous Positive Airway Pressure (CPAP), Non-Invasive Neurally Adjusted Ventilatory Assist (NIV-NAVA), Non-Invasive Ventilator (NIV), High Flow Nasal Cannula (>2L), and Non-invasive positive pressure ventilation (NIPPV)

Exclusion Criteria:

* Infants participating in other music therapy studies.
* Infants in custody of Children's Division
* Requiring non-invasive respiratory support that does not inhibit the start of oral feeding, including High Flow Nasal Cannula (≤ 2L), Nasal Cannula
* Requiring no respiratory support
* Requiring invasive respiratory support
* Infants who are diagnosed with congenital malformations of bowel or bowel perforations
* Infants diagnosed with surgical necrotizing enterocolitis

Ages: 1 Day to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Oral Feeding | 1-6 weeks
  Time to full transition from gavage to oral feeding by mouth as measured by days

SECONDARY OUTCOMES:
Length of Stay | 1-8 months
  Length of time admitted in the NICU as measured by days
Length of Respiratory Support | 1-16 weeks
  Length of time before transition to breathing room air as measured by days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri Healthcare, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
We have no plan to make IPD available to other researchers.

REFERENCES:
- [Background] Dumpa V, Kamity R, Ferrara L, Akerman M, Hanna N. The effects of oral feeding while on nasal continuous positive airway pressure (NCPAP) in preterm infants. J Perinatol. 2020 Jun;40(6):909-915. doi: 10.1038/s41372-020-0632-2. Epub 2020 Feb 21. PMID 32086439
- [Background] Chorna OD, Slaughter JC, Wang L, Stark AR, Maitre NL. A pacifier-activated music player with mother's voice improves oral feeding in preterm infants. Pediatrics. 2014 Mar;133(3):462-8. doi: 10.1542/peds.2013-2547. Epub 2014 Feb 17. PMID 24534413
- [Background] Glackin SJ, O'Sullivan A, George S, Semberova J, Miletin J. High flow nasal cannula versus NCPAP, duration to full oral feeds in preterm infants: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2017 Jul;102(4):F329-F332. doi: 10.1136/archdischild-2016-311388. Epub 2016 Dec 23. PMID 28011792
- [Background] Hanin M, Nuthakki S, Malkar MB, Jadcherla SR. Safety and Efficacy of Oral Feeding in Infants with BPD on Nasal CPAP. Dysphagia. 2015 Apr;30(2):121-7. doi: 10.1007/s00455-014-9586-x. Epub 2014 Nov 8. PMID 25380678
- [Background] Hatch LD 3rd, Clark RH, Carlo WA, Stark AR, Ely EW, Patrick SW. Changes in Use of Respiratory Support for Preterm Infants in the US, 2008-2018. JAMA Pediatr. 2021 Oct 1;175(10):1017-1024. doi: 10.1001/jamapediatrics.2021.1921. PMID 34228110
- [Background] Jain D, Bancalari E. New Developments in Respiratory Support for Preterm Infants. Am J Perinatol. 2019 Jul;36(S 02):S13-S17. doi: 10.1055/s-0039-1691817. Epub 2019 Jun 25. PMID 31238352